CLINICAL TRIAL: NCT00039091
Title: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 (Anti-CTLA-4) Humanized Monoclonal Antibody (MDX-CTLA-4 NSC# 732442, Previously 720801) in Patients Previously Vaccinated With GM-CSF-Based Autologous Tumor Vaccines (CTEP Protocol Number P-5708) and Patients With Acute Myelogenous Leukemia/ Myelodysplasia, and Non-Small Cell Lung Cancer Who Have Not Received a Prior Vaccine
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Ovarian Epithelial Cancer, Melanoma, Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03144; 01-228; R21CA105776 (NIH); CDR0000069349 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Melanoma; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Stage IV Melanoma; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myeloid, Acute; Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial | interventions — Ipilimumab; CTLA-4 Antigen

ARMS (1):
- Treatment (ipilimumab) (Experimental): Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody IV over 90 minutes on day 1. Courses repeat every 2 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ipilimumab

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4

SUMMARY:
This phase I trial is studying the side effects of monoclonal antibody therapy in treating patients with ovarian epithelial cancer, melanoma, acute myeloid leukemia, myelodysplastic syndrome, or non-small cell lung cancer. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of MDX-CTLA-4 in patients previously and not previously vaccinated with GM-CSF-based vaccines using lethally irradiated, autologous melanoma, ovarian cancer, acute myelogenous leukemia/myelodysplasia or lung cancer cells.

II. To identify preliminary evidence of biologic activity and efficacy.

OUTLINE:

Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody IV over 90 minutes on day 1. Courses repeat every 2 months in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly until disease progression.

PROJECTED ACCRUAL: A total of 48 patients (12 per disease type; 36 previously treated with a sargramostim (GM-CSF)-expressing autologous tumor cell vaccine and 12 not previously treated with this vaccine) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously vaccinated with GM-CSF-based vaccines using lethally irradiated, autologous melanoma, ovarian cancer, acute myelogenous leukemia/myelodysplasia, or non-small cell lung cancer cells; patients with acute myelogenous leukemia/myelodysplasia or non-small cell lung cancer who have not been vaccinated with an autologous, GM-CSF based vaccine
* >= 4 weeks since treatment (chemo-, radiation, hormone, immuno-, etc., therapy)
* Patients must have recovered from any acute toxicity associated with prior therapy
* Measurable epithelial ovarian cancer, melanoma, AML/MDS, or non-small cell lung cancer
* No standard curative treatment options
* Not require immediate palliative therapy
* Patients with epithelial ovarian cancer must have persistent or recurrent disease following primary surgery and primary chemotherapy
* Patients with melanoma must be stage IV disease
* Patients with AML/MDS, but without MDS, must be: a) in second relapse or b) first relapse with no option for bone marrow transplant or c) not a candidate for immunosuppressive chemotherapy due to age or comorbid disease
* Patients with non-small cell lung cancer must be not curable by standard surgery, chemotherapy, and/or radiation
* Life expectancy >= 12 weeks
* ECOG performance status of 0, 1 or 2
* Written informed consent
* Due to the unknown effects of MDX-CTLA-4 on the fetus or nursing infant, pregnant or nursing women should not be included; women should be either: post-menopausal for at least 1 year; surgically incapable of bearing children; or utilizing an intrauterine device, and/or spermicide and barrier, for contraception; during the study, use of oral contraception alone is not acceptable; women of childbearing potential must have a negative serum beta-HCG pregnancy test conducted during screening, and a negative urinary beta-HCG pregnancy test conducted within 24 hours prior to treatment; due to the unknown effects of MDX-CTLA-4 on the fetus, men should not father children during the study
* WBC > 1,000 cells/mm^3 (except for AML/MDS patients)
* Serum creatinine < 2 mg/dL
* Platelets > 75,000 cells/mm^3 (except for AML/MDS patients)
* AST and ALT < 2 x UNL
* Total bilirubin < 2 x UNL

Exclusion Criteria:

* Active infection
* Autoimmune disease requiring immunosuppressive treatment
* Any underlying medical condition which, in the principal investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* Any concurrent medical condition requiring the use of systemic steroids (use of inhaled or topical steroids is acceptable)
* CNS metastases, unless previously treated and stable for at least three months
* Patients who have received prior treatment with MDX-CTLA-4

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11-21 (Actual)

PRIMARY OUTCOMES:
Toxicities of ipilimumab, based on the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 6 years

SECONDARY OUTCOMES:
Overall clinical response rate (complete response [CR] plus partial response [PR]) based on the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 years
  90% confidence intervals will be estimated.
Proportion of patients who mount a brisk immune response, graded as absent, non-brisk, and brisk as described by Mihm | Up to 2 months post-treatment
  90% confidence intervals will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hodi, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States